CLINICAL TRIAL: NCT00349674
Title: Treatment of ANCA-Associated Vasculitides : Corticosteroids and Pulse Cyclophosphamide Followed by Maintenance Therapy With Methotrexate or Azathioprine: a Prospective Multicenter Randomized Trial
Brief Title: WEGENT - Comparison of Methotrexate or Azathioprine as Maintenance Therapy for ANCA-Associated Vasculitides
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 97.129
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Systemic Wegener's Granulomatosis
Keywords: Wegener's granulomatosis,; microscopic polyangiitis,; ANCA-associated vasculitis,; methotrexate,; azathioprine
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Azathioprine; Methotrexate

INTERVENTIONS:
Drug: Azathioprine: 2 mg/kg/day
Drug: methotrexate 0.3 mg/kg/week, to a maximum and optimal dose of 25 mg/week

SUMMARY:
Remission of ANCA-associated vasculitis can be obtained in approximately 80% of the patients with a combination of corticosteroids and cyclophosphamide. However, relapses are frequent. This point warrants the prescription of a maintenance treatment with a less toxic immunosuppressant for several months to years. The optimal drug in this indication is not determine. We decided therefore to compare the 2 most used drugs in this indication. Induction therapy consists in the combination of corticosteroids and intravenous cyclophosphamide pulses. Corticotherapy consisted first in one daily methylprednisolone pulse, for 1 to 3 days, followed by oral prednisolone at the dose of 1 mg/kg/d for 3 weeks, then progressively tapered and stopped at the 18th month from the diagnosis. Cyclophosphamide is administered every 2 weeks for the first 3 bolus (0.6 g/m2 - D1, 15 and 30), then every 3 weeks (0.7 g/m2). Once remission is achieved, patients receive 3 additional bolus (0.7 g/m2). At that time, patients are randomized for a maintenance treatment with azathioprine (2 mg/kg/d, orally) or oral methotrexate (starting at the dose of 0.3 mg/kg/wk, then progressively increased every weeks by 2.5mg, if necessary, to a maximum and optimal dose of 25 mg/wk) for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years-old with newly diagnosed systemic Wegener's granulomatosis,
* microscopic polyangitis with at least one factor of poor prognosis according to the five factors score (proteinuria > 1 g/day, renal insufficiency defined as a serum creatininemia > 140 µmol/L, specific cardiomyopathy, gastrointestinal tract and/or CNS involvement).

Exclusion Criteria:

* MPA patients with no poor prognosis factor;
* localized WG;
* relapse of previously known WG or MPA;
* treatment with corticosteroids for more than 1 month prior to diagnosis and start of immunosuppressant;
* co-existence of another multi-system autoimmune disease;
* malignancy (unless considered in complete remission and with no therapy for at least 3 years);
* contra-indication to corticosteroids or study immunosuppressants; pregnancy or no use of contraception in non-menopaused women;
* infection with human immunodeficiency virus; mental or physical disturbances not permitting to give consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126
Dates: Start 1999-01

PRIMARY OUTCOMES:
Safety/Efficacy
Frequency of severe adverse events in each arm. Hypothesis based upon NIH data was a rate of 6% severe adverse event with methotrexate compared to 30% with azathioprine (24% in one study on RA and 46% in one study on Sjögren syndrome).
Evaluation was planned after the last included patient has completed the assigned trial regimen (after 12 months of maintenance regimen or because of drug withdrawal).

SECONDARY OUTCOMES:
Relapse-free survival rate.
Cumulative event-free survival rate (adverse event- and relapse-free survival rate).
Health quality assessment using HAQ and SF36.
Efficacy of induction therapy with pulsed cyclophosphamide.
Second evaluation of the same outcome parameters is planned 5 years after the last included patient has completed the assigned trial regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François CORDIER, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Christian PAGNOUX, Paris, France

REFERENCES:
- [Derived] Pagnoux C, Mahr A, Hamidou MA, Boffa JJ, Ruivard M, Ducroix JP, Kyndt X, Lifermann F, Papo T, Lambert M, Le Noach J, Khellaf M, Merrien D, Puechal X, Vinzio S, Cohen P, Mouthon L, Cordier JF, Guillevin L; French Vasculitis Study Group. Azathioprine or methotrexate maintenance for ANCA-associated vasculitis. N Engl J Med. 2008 Dec 25;359(26):2790-803. doi: 10.1056/NEJMoa0802311. PMID 19109574